CLINICAL TRIAL: NCT03868085
Title: The Natural History of Injury-Related Disuse Osteopenia
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, J. Spence Reid, Professor and Chief, Division of Orthopaedic Trauma, Milton S. Hershey Medical Center
Other Study IDs: 00006601
Record Dates: First submitted 2017-05-30; First posted 2019-03-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: dual energy x-ray absorptiometry — DXA scan

SUMMARY:
Determine the severity and time course (natural history) of disuse osteopenia that occurs in the lower extremity(ies) and lumbar spine of patients sustaining lower extremity injuries that require the patient to maintain restricted weight bearing status (12 weeks) following the surgical fixation of the patient's injuries.

The investigators hypothesize that there will be a significant decrease in the bone mineral density in the lower limbs of patients undergoing restricted weight bearing for peri-articular injuries of the lower extremity. This loss of bone mineral density is often prolonged in its duration and may lower subsequent fracture threshold and prolong the time to recovery and return to activities.

DETAILED DESCRIPTION:
It is well documented that restricted weight bearing even for relatively short periods (12 weeks) associated with the surgical treatment of peri-articular injuries of the lower extremity (ie acetabulum, distal femur, tibial plateau, pilon, talus, calcaneus) can lead to a measurable decrease in bone density in the injured limb. Furthermore, this osteopenia can persist for extended periods of time - much longer than the original period of restricted weight bearing. This relative osteopenia can delay recovery from injury, lower fracture threshold for subsequent injury and potentially delay return to active duty in the case of a wounded warrior. There exists a significant body of research in the modulation of the osteopenia associated with restricted weight bearing as it pertains to long term space flight (microgravity).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 at time of injury
2. Previously normal community ambulator (without ambulatory aid) prior to injury

Exclusion Criteria:

1. Presence of a total or hemi hip prosthesis in the injured extremity
2. Presence of lumbar fusion L1-L4
3. Previous ipsilateral lower extremity trauma
4. History of medical treatment for known osteoporosis (Calcium and Vitamin D supplementation alone is NOT an exclusion criteria)
5. Ambulatory dysfunction prior to injury
6. Inability to cooperate with DXA scanning
7. Head injury on admission requiring invasive monitoring or treatment
8. Inability to adhere to weight bearing restrictions
9. Inability to provide consent
10. Non English speaking
11. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Patients with one or more of the following lower extremity peri-articular fractures with restricted weight bearing for 12 weeks: (OTA types A,B,C). Injuries may be unilateral or bilateral.
  1. Acetabulum fracture
  2. Distal Femur fracture
  3. Tibial plateau fracture
  4. Pilon fracture
  5. Talus fracture
  6. Calcaneus fracture
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Determine the natural history of disuse osteopenia following restricted weight bearing from a lower extremity articular injury | 36 months
  Hip bone mineral density (DXA) of control and injured limb will be measured following weight bearing restrictions as part of treatment of lower limb articular injury and again following resumption of weight bearing after healing of the injury.

CONTACTS AND LOCATIONS:
Overall Officials: John S Reid, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No